CLINICAL TRIAL: NCT00493831
Title: Analysis of Lipid Biomarkers of Exposure and Host Response
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: primary analyses found futile
Sponsor: University of Nebraska (Other)
Collaborators: Lorillard Tobacco Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0256-05-FB
Record Dates: First submitted 2007-06-05; First posted 2007-06-28 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Cigarette Smoking
Keywords: smoking reduction; inflammation; harm reduction; lipid biomarkers
MeSH Terms: conditions — Cigarette Smoking; Smoking Reduction; Inflammation; Harm Reduction | interventions — Tobacco Use Cessation Devices; Transdermal Patch; Nebulizers and Vaporizers; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine replacement therapy (NRT) (Experimental): any form of nicotine replacement would be allowed at subject discretion
  Interventions: Drug: nicotine polacrilex, transdermal system or inhaler

INTERVENTIONS:
Drug: nicotine polacrilex, transdermal system or inhaler — on label use of Nicotine replacement therapy (NRT)
  Other Names: Nicotine replacement therapy

SUMMARY:
The purpose of this prospective, open-label, clinical trial is to establish the feasibility and validity of exhaled breath condensate (EBC) biomarkers for use in studies designed to evaluate harm reduction strategies of smoking. This will be accomplished by measuring selected markers in EBC believed related to the pathogenesis of lung disease before and after a smoking cessation intervention.

DETAILED DESCRIPTION:
Twenty subjects will be accrued in three groups based on smoking habit: 10-20, 20-30 and >30 cigarettes/day. Eligibility criteria include male and female cigarette smokers ≥19 years of age, who are able to give informed consent, able to exhale into Eco Screen instrument for 15-20 minutes. All must be willing to make a serious quit attempt and be willing to use nicotine replacement therapy.

Subjects will be excluded if any of the following are present: regular use of anti-inflammatory medication; presence of any inflammatory disease of the respiratory tract including moderate or worse COPD (FEV1 < 80% predicted and FEV1/FVC ratio < 0.7). Subjects with normal lung function who meet criteria for diagnosis of chronic bronchitis will be excluded. Subjects with stable medical conditions, excluding inflammatory lung disease, will be permitted to participate, providing anti-inflammatory therapies are not used regularly and providing there has been no change in their clinical status in the two months prior to beginning the study.

Upon entering into the study, subjects will establish a quit date and will be treated with nicotine replacement therapy (NRT) products based on individual preference and will receive smoking cessation counseling. They will then be seen at 12 visits over the course of 25 weeks.

Evaluations will include vital signs, interval smoking history, food frequency questionnaire, exhaled carbon monoxide, blood drawn for chemistry and CBC, peripheral blood harvested and serum aliquoted and saved for future biochemical analysis, urine sample for isoprostane, pregnancy test for females, and exhaled breath condensate. Some visits may also include spirometry with and with out bronchodilators, 24 hour urine collections for NNAL and NNAL-glc quantification, health status assessed using St. George's Respiratory Questionnaire, the Functional Assessment of Chronic Illness Therapy - Fatigue, the Leicester Cough Questionnaire, the Clinical COPD Questionnaire and smoking related symptoms assessed using the Breathlessness, Cough, and Sputum Scale.

ELIGIBILITY:
Inclusion Criteria:

* Smoke at least 5 pack years
* Have a stable smoking habit for 3 months
* Be willing to make a serious quit attempt and
* Be able to use nicotine replacement therapy

Exclusion Criteria:

* Regular use of an anti-inflammatory medication
* Presence of an inflammatory lung disease
* Unstable medical condition

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-08-23 (Actual); Primary Completion 2007-09-09 (Actual); Study Completion 2007-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen I Rennard, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 subjects were recruited, but only 20 proceeded to the intervention. Some information was collected from all 20, although outcomes were not measurable in any.
Groups:
- Nicotine Replacement Therapy: open label self comparison study design
  nicotine polacrilex, transdermal system or inhaler
Period: Overall Study
Arm/Group | Nicotine Replacement Therapy
Started | 20 (24 subjects were consented but only 20 continued to the treatment phase. Of these 12 completed. The study was terminated as the analyses proved infeasible prior to the other subjects completed)
Completed | 12
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Study terminated as primary analysis not feasible; the number of 24 included in the analysis population was based on subjects consented. No analyses were successfully done. Baseline was defined as before intervention, and is listed as 20 as only 20 subjects entered the treatment phase.
Units Other Than Participants: number
Groups:
- Nicotine Replacement Therapy: any form of nicotine replacement would be allowed at subject discretion
  nicotine polacrilex, transdermal system or inhaler: on label use of NRT
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 20
Number analyzed (number) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Lipid Measures in EBC
Description: No data were collected
Time Frame: 12 weeks
Population: Study withdrawn so no data available for analysis. No data collected.
Arm/Group | Nicotine Replacement Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study withdrawn
Description: Study withdrawn
Arm/Group | Nicotine Replacement Therapy
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
The exhaled breath condensates did not contain sufficient lipids to permit evaluation above limits of detectability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No